CLINICAL TRIAL: NCT07017062
Title: Clinical Evaluation of Hybrid Ceramic Occlusal Veneers Bonded With Two Self Adhesive Resin Cements A Randomized Clinical Trial
Brief Title: Clinical Evaluation of Hybrid Ceramic Occlusal Veneers Bonded With Two Self Adhesive Resin Cements
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Hayat Ibrahim Mahrous Ibrahim, principal investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2010777
Record Dates: First submitted 2025-05-31; First posted 2025-06-12 (Actual); Last update posted 2025-06-12 (Actual); Status verified 2025-06

CONDITIONS: Occlusal Wear of Teeth

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Hybrid ceramic occlusal veneers cemented with Rely X U200 cement (Active Comparator)
  Interventions: Other: hybrid ceramic occlusal veneers
- Hybrid ceramic occlusal veneers cemented with BeautiLink SA cement (Experimental)
  Interventions: Other: hybrid ceramic occlusal veneers

INTERVENTIONS:
Other: hybrid ceramic occlusal veneers — occlusal veneers cemented with self adhesive resin cements

SUMMARY:
This randomized clinical trial aims to evaluate the clinical performance of hybrid ceramic occlusal veneers cemented with two different bonding protocols: a self-adhesive bonding protocol with adhesive enhancement (BeautiLink SA cement with BeautiBond Xtreme adhesive) versus another self-adhesive bonding protocol (RelyX U200 self-adhesive resin cement with 3M UNIVERSAL bond).

ELIGIBILITY:
Inclusion Criteria:

* • Age ≥ 21 years

  * Vital teeth
  * Sufficient tooth structure for veneer retention
  * Willing and able to provide written informed consent
  * Ability to attend all follow-up appointments
  * Adequate oral hygiene as determined by the investigator

Exclusion Criteria:

* • Patients with active periodontal disease (probing depth > 4mm, bleeding on probing)

  * Patients with severe parafunctional habits (e.g., bruxism confirmed by clinical examination)
  * Poor oral hygiene (plaque index > 30%)
  * Pregnancy or nursing
  * Systemic diseases affecting treatment outcomes (e.g., uncontrolled diabetes, immunosuppression)
  * Known allergies to study materials (ceramic, or resin cement components)
  * Inability to comply with study requirements
  * Current participation in other dental clinical trials
  * Active orthodontic treatment

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2025-06 (Estimated); Primary Completion 2025-07 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Marginal discoloration | 18 months
  Measuring device: Modified USPHS criteria Alpha: No discoloration on margin Bravo: Discoloration found at margin Charlie: Discoloration with penetration in a pulpal direction

SECONDARY OUTCOMES:
Retention | 18 months
  Measuring device: Modified USPHS criteria Alpha: retained Charlie: debonded
Marginal adaptation | 18 months
  Measuring device: Modified USPHS criteria Alpha: explorer does not catch or has one way catch when drawn across restoration/tooth interface Bravo: explorer falls into crevice when drawn across the restoration tooth interface Charlie: Dentin or base exposed along margin
Postoperative hypersensitivity | 18 months
  Measuring device: Modified USPHS criteria Alpha: Absent Charlie: Present
Recurrent caries | 18 months
  Measuring device: Modified USPHS criteria Alpha: no evidence of caries at the margin of restoration Charlie: evidence of caries continuous with the margin of restoration

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Dentistry, Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided